CLINICAL TRIAL: NCT06602414
Title: Is Conservative Treatment Still an Option for Distal Biceps Tendon Lesions? Evaluation of Clinical Results of Patients Treated Conservatively for Distal Biceps Tendon Lesions at 1 Year Minimum Follow-up
Brief Title: Evaluation of Clinical Results of Patients Treated Conservatively for Distal Biceps Tendon Lesions
Acronym: CoB
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 340/2024/Oss/IOR
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Tendon Rupture
Keywords: Distal Biceps tendon rupture; Elbow tendon ruptures; Elbow tendon ruptures conservative treatment
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Conservative treatment: Patients treated conservatively for distal biceps tendon rupture
  Interventions: Procedure: Conservative treatment

INTERVENTIONS:
Procedure: Conservative treatment — Conservative treatment instead of surgical repair

SUMMARY:
A clinical evaluation of the results of conservative treatment after distal biceps tendon rupture with a minimum follow up of 1 year.

The results will be evaluated with clinical scores (MEPS, DASH and SF-12) and strenght and fatigue evaluations with dynamometers for both flexion and supination of elbow and forearm. The results of the affected side will be compared with the controlateral side

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old at time of injury
* Complete acute distal biceps tendon rupture diagnosed and evaluated at IRCCS Istituto ortopedico Rizzoli between 2000 and 2024 treated conservatively

Exclusion Criteria:

* < 18 years at time of injury
* Patients who present controindications to the strenght evaluation
* Patients who have developed other non correlated injuries to the affected arm (e.g. fractures or tendon injuries)
* Patients treated surgically for distal biceps tendon rupture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have suffered an acute distal biceps tendon rupture
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Elbow Function | At baseline (day 0)
  The Mayo Elbow Performance score (MEPS) or Mayo Elbow Performance Index (MEPI) is an instrument used to test the limitations, caused by pathology, of the elbow during activities of daily living (ADL) . This specific test uses 4 subscales:
  Pain, Range of Motion (arc of motion of the art. humeroulnaris) Stability Daily Function MEPS can be used to measure which treatment work best for different conditions, An example would be when deciding the best post-operative treatment for example: the difference in prognosis between open and closed fractures when operated.
  This numerical scale express results on a scale from 0 to 100 and considers results with a score higher than 85 as excellent results.

SECONDARY OUTCOMES:
Upper Limb Function | At baseline (day 0)
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale.
  The QuickDASH is an abbreviated version of the original DASH outcome measure. In comparison to the original 30 item DASH outcome measure, the QuickDASH only contains 11 items It is a questionnaire that measures an individual's ability to complete tasks, absorb forces, and severity of symptoms. The QuickDASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity/function level.
  The DASH score expresses results on a scale from 0 to 100 with 0 considered as no disabilities and 100 as maximum disability.
Short Form Health Survey | At baseline (day 0)
  The Short Form (12) Health Survey is a 12-item, patient-reported survey of patient health. It is a reduced size version of the SF-36, and is widely used since it produces similar results for physical and mental health scores with far less respondent burden for producing scores of overall mental and physical well-being.
  The mean score obtained by the US population is 50 points, any differentiation of 10 points represents a difference of 1 standard deviation from the mean values.
Flexion strenght | At baseline (day 0)
  Measured with dynamometer considering the maximum value obtained out of 10 repetition, expressed in Kg.
Flexion Fatigue | At baseline (day 0)
  Measuring the difference of strenght between the first and final pull of a series of 10 repetitions. Expressed in Kg
Supination Strenght | At baseline (day 0)
  Measured with dynamometer considering the maximum value obtained out of 10 repetition, expressed in Kg.
Supination Fatigue | At baseline (day 0)
  Measuring the difference of strenght between the first and final pull of a series of 10 repetitions. Expressed in Kg

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

REFERENCES:
- [Background] Srinivasan RC, Pederson WC, Morrey BF. Distal Biceps Tendon Repair and Reconstruction. J Hand Surg Am. 2020 Jan;45(1):48-56. doi: 10.1016/j.jhsa.2019.09.014. PMID 31901332
- [Background] Athwal GS, Steinmann SP, Rispoli DM. The distal biceps tendon: footprint and relevant clinical anatomy. J Hand Surg Am. 2007 Oct;32(8):1225-9. doi: 10.1016/j.jhsa.2007.05.027. PMID 17923307